CLINICAL TRIAL: NCT02401152
Title: The Effect of a Potato Based Low-osmolaric Glucose Polymer Drink on Gastric Distress and Running Performance
Brief Title: A Low-osmolaric Glucose Polymer Drink for Gastric Distress and Running Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoSportNL (Other)
Collaborators: Avebe U.A. (Unknown)
Responsible Party: Principal Investigator, Jeroen Wouters, Dr. Ir., InnoSportNL
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: LOGP-001
Record Dates: First submitted 2015-03-09; First posted 2015-03-27 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Gastric Distress; Running Performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo group (Placebo Comparator): Sports drink containing maltodextrin
  Interventions: Other: Placebo
- Sports drink 1 (Active Comparator): Sports drink with a specific source of carbohydrates (CHO).
  Interventions: Other: Sports drink 1
- Sports drink 2 (Active Comparator): Sports drink with a specific source of CHO.
  Interventions: Other: Sports drink 2

INTERVENTIONS:
Other: Sports drink 1 — Sports drink with a specific source of CHO.
  Arms: Sports drink 1
Other: Sports drink 2 — Sports drink with a specific source of CHO
  Arms: Sports drink 2
Other: Placebo — iso-caloric sports drink with maltodextrin as CHO source
  Arms: Placebo group

SUMMARY:
The objective of this study is to investigate whether two newly developed sports drink will affect gastric distress (GD) and running performance (RP) compared to an iso-caloric control drink both in a short and longer distance run. Furthermore, the effect of the newly developed sports drinks on gastric emptying will be investigated.

The study will consist of 3 parts. Firstly, a randomized cross-over design is used for the short distance run and the effects on GD and RP. Secondly, a parallel design is used to study the effects of the drinks on GD and RP during a longer distance run. Thirdly, the gastric emptying tests will be performed in a randomized cross-over design. Participants will be asked to fill in questionnaire on the gastric distress they experience. 40 participants will be enrolled to participate in part 1 and part 2. 10 out of 40 will participate in part 3 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* A BMI between 18.5 and 25 kg*m-2
* Intermediate level runners with at least 1 year of running experience, performing moderate to intensive running exercise consistently (two or more times per week for a minimum of 30 minutes each time)

Exclusion Criteria:

* Pregnancy
* Having diseases, such as diabetes, kidney, liver, lung, or bowel disease, cardiovascular disease, or mental illness
* Abuse of alcohol (>20 alcoholic consumptions per week)
* Use of medication and/or drugs
* Smoking/having smoked in the last six months
* Participating in any scientific intervention providing a treatment potentially interfering with this study's treatment (to be decided by the researchers)
* Allergic to one of the components present in the drinks, including milk (incl. lactose), soy and gluten

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Perceived degree of gastric complaints after consumption of sports drink and running exercise | Approximately 10-20 minutes for the 3 km and 40-60 minutes for the 10 km.
  Quantified as the score for the perceived degree of experiencing 7 different gastric complaints on a VAS. The total score for gastric distress and the scores for each different gastric complaint will be analysed separately for the three different time points (before, during and after exercise). The total score is the sum of the scores on the separate complaints.
Finishing time during 10 km running event | Depending on the speed of the participant, an average time frame of 40-60 minutes after starting the run is expected.

SECONDARY OUTCOMES:
Rate of gastric emptying | 1 hour after ingestion of sports drink
  During 1 hour after ingestion of the sports drink, subjects will breath into a specific bag which will be analysed for the presence of C13 on specific time points. The decrease of C13 in the exhaled air is a measurement for gastric emptying time.
Blood glucose levels | During 1 hour after ingestion of sports drink
  On specific time points within 1 hour after ingestion of the sports drink, blood glucose levels will be determined to calculate area under the curve for the different sport drinks.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Wouters, Dr. Ir., Principal Investigator
Locations (1):
- InnoSportlab Papendal, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Background] Leiper JB, Aulin KP, Soderlund K. Improved gastric emptying rate in humans of a unique glucose polymer with gel-forming properties. Scand J Gastroenterol. 2000 Nov;35(11):1143-9. doi: 10.1080/003655200750056600. PMID 11145284
- [Background] Takii H, Takii Nagao Y, Kometani T, Nishimura T, Nakae T, Kuriki T, Fushiki T. Fluids containing a highly branched cyclic dextrin influence the gastric emptying rate. Int J Sports Med. 2005 May;26(4):314-9. doi: 10.1055/s-2004-820999. PMID 15900642
- [Background] Stephens FB, Roig M, Armstrong G, Greenhaff PL. Post-exercise ingestion of a unique, high molecular weight glucose polymer solution improves performance during a subsequent bout of cycling exercise. J Sports Sci. 2008 Jan 15;26(2):149-54. doi: 10.1080/02640410701361548. PMID 17852670
- [Background] Rehrer NJ, Brouns F, Beckers EJ, ten Hoor F, Saris WH. Gastric emptying with repeated drinking during running and bicycling. Int J Sports Med. 1990 Jun;11(3):238-43. doi: 10.1055/s-2007-1024799. PMID 2373584
- [Background] Moses FM. The effect of exercise on the gastrointestinal tract. Sports Med. 1990 Mar;9(3):159-72. doi: 10.2165/00007256-199009030-00004. PMID 2180030
- [Background] de Oliveira EP, Burini RC. Food-dependent, exercise-induced gastrointestinal distress. J Int Soc Sports Nutr. 2011 Sep 28;8:12. doi: 10.1186/1550-2783-8-12. PMID 21955383
- [Background] Ploutz-Snyder L, Foley J, Ploutz-Snyder R, Kanaley J, Sagendorf K, Meyer R. Gastric gas and fluid emptying assessed by magnetic resonance imaging. Eur J Appl Physiol Occup Physiol. 1999 Feb;79(3):212-20. doi: 10.1007/s004210050498. PMID 10048625
- [Background] Rodriguez NR, DiMarco NM, Langley S; American Dietetic Association; Dietitians of Canada; American College of Sports Medicine: Nutrition and Athletic Performance. Position of the American Dietetic Association, Dietitians of Canada, and the American College of Sports Medicine: Nutrition and athletic performance. J Am Diet Assoc. 2009 Mar;109(3):509-27. doi: 10.1016/j.jada.2009.01.005. PMID 19278045
- [Background] American Dietetic Association; Dietitians of Canada; American College of Sports Medicine; Rodriguez NR, Di Marco NM, Langley S. American College of Sports Medicine position stand. Nutrition and athletic performance. Med Sci Sports Exerc. 2009 Mar;41(3):709-31. doi: 10.1249/MSS.0b013e31890eb86. PMID 19225360
- [Background] Murray R, Bartoli W, Stofan J, Horn M, Eddy D. A comparison of the gastric emptying characteristics of selected sports drinks. Int J Sport Nutr. 1999 Sep;9(3):263-74. doi: 10.1123/ijsn.9.3.263. PMID 10477362
- [Background] Maughan RJ, Leiper JB. Limitations to fluid replacement during exercise. Can J Appl Physiol. 1999 Apr;24(2):173-87. doi: 10.1139/h99-015. PMID 10198143
- [Background] Rowlands DS, Wallis GA, Shaw C, Jentjens RL, Jeukendrup AE. Glucose polymer molecular weight does not affect exogenous carbohydrate oxidation. Med Sci Sports Exerc. 2005 Sep;37(9):1510-6. doi: 10.1249/01.mss.0000177586.68399.f5. PMID 16177602
- [Background] Zhu Y, Hsu WH, Hollis JH. The impact of food viscosity on eating rate, subjective appetite, glycemic response and gastric emptying rate. PLoS One. 2013 Jun 20;8(6):e67482. doi: 10.1371/journal.pone.0067482. Print 2013. PMID 23818981
- [Background] Siegel JA, Krevsky B, Maurer AH, Charkes ND, Fisher RS, Malmud LS. Scintigraphic evaluation of gastric emptying: are radiolabeled solids necessary? Clin Nucl Med. 1989 Jan;14(1):40-6. doi: 10.1097/00003072-198901000-00011. PMID 2714039
- [Background] Chang TM, Passaro E Jr, Shain LR, Chen WL. Physical properties of starch meals in vivo and in vitro and their influence on gastric emptying and oral glucose tolerance test. Nutrition. 1991 Nov-Dec;7(6):410-6. PMID 1802230
- [Background] Mourot J, Thouvenot P, Couet C, Antoine JM, Krobicka A, Debry G. Relationship between the rate of gastric emptying and glucose and insulin responses to starchy foods in young healthy adults. Am J Clin Nutr. 1988 Oct;48(4):1035-40. doi: 10.1093/ajcn/48.4.1035. PMID 3048076